CLINICAL TRIAL: NCT05868252
Title: Molecular Analysis of Screen Detected Non-invasive Breast Cancer and Atypical Breast Hyperplasias Identified by the Sloane Project
Brief Title: Molecular Analysis of the Sloane Project
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19/LO/0648
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: DCIS; LCIS; Atypical Ductal Hyperplasia; Atypical Lobular Hyperplasia
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Sloane Project is a UK wide prospective audit of screen detected non-invasive and atypical breast hyperplasias named after John Sloane an eminent pathologist interested in the field. Non invasive breast neoplasia accounts for 25% of all 'breast cancers' detected through breast screening and includes ductal carcinoma in situ (DCIS) and lobular carcinoma in situ (LCIS). Atypical hyperplasias are high risk but benign lesions found in 10% of benign biopsies performed through the NHS breast screening programme. The importance of these lesions rests on the increased risk of subsequently developing invasive breast cancer, with DCIS at highest risk (20 times greater than the general population) followed by LCIS (10 times greater) and atypical breast hyperplasia (4 times greater).

The Sloane Project data are held by Public Health England (PHE) and provide full and detailed information about the patients' journey from diagnosis to treatment and outcome. The project aims to increase the understanding of how best to manage these early lesions which can lead to breast cancer.

All NHS breast screening units in the UK are invited to submit data for the Sloane Project. Historically an exceptional ~90% of centres in England, Scotland, Wales and Northern Ireland have participated on a voluntary basis.

The objective of this research protocol is the collection of anonymised formalin fixed paraffin embedded (FFPE) tissue blocks from women whose data is held within the Sloane Project database in order to allow detailed analysis of the biological, molecular and genomic changes in these cases of in situ carcinoma and atypical hyperplasia and how these relate to the corresponding annotated clinical, pathological and radiological data already collected by and held in PHE. We seek to identify particular signature(s) that define which patients are likely to develop invasive disease, distinguishing the worrisome from indolent, non-worrisome lesions.

ELIGIBILITY:
Inclusion Criteria:

* DCIS (Ductal Carcinoma in situ)
* LCIS (Lobular Carcinoma in situ)
* Atypical hyperplasias

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Those who have undergone breast screening and were part of the Sloane Project audit
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-05-19 (Estimated); Study Completion 2024-05-19 (Estimated)

PRIMARY OUTCOMES:
Progression of breast disease | From diagnosis to end of 2016

CONTACTS AND LOCATIONS:
Overall Officials: Elinor Sawyer, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No